CLINICAL TRIAL: NCT01905150
Title: Ph 2 Trial of G-FLIP (Low Doses Gemcitabine, 5FU, Leucovorin, Irinotecan & Oxaliplatin), Followed by G-FLIP-DM (G-FLIP + Low Doses Docetaxel & MitomycinC), When Used in Combination With Vitamin C, in Patients With Advanced Pancreatic Cancer
Brief Title: Ph 2 Trial of Vitamin C & G-FLIP (Low Doses Gemcitabine, 5FU, Leucovorin, Irinotecan, Oxaliplatin) for Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bruckner Oncology (Other)
Collaborators: Hirschfeld Oncology (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 119005
Record Dates: First submitted 2013-07-18; First posted 2013-07-23 (Estimated); Results first posted 2024-08-14 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2020-01

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic Cancer; G-FLIP, Gemcitabine 5FU Leucovorin Irinotecan Oxaliplatin; G-FLIP-DM (G-FLIP + Low doses Docetaxel and Mitomycin C); Vitamin C (ascorbic acid)
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Fluorouracil; Leucovorin; Irinotecan; Oxaliplatin; Gemcitabine; Docetaxel; Mitomycin; Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- G-FLIP+VitaminC, then G-FLIP-DM+VitaminC (Experimental): G-FLIP in combination with Vitamin C, then G-FLIP-DM in combination with Vitamin C
  Interventions: Drug: G-FLIP; Drug: G-FLIP-DM; Dietary Supplement: Vitamin C
- G-FLIP, then G-FLIP-DM (Active Comparator): G-FLIP alone, then G-GLIP-DM alone
  Interventions: Drug: G-FLIP; Drug: G-FLIP-DM

INTERVENTIONS:
Drug: G-FLIP — G-FLIP is a combination of Low Doses of Gemcitabine, Fluorouracil [5FU], Leucovorin, Irinotecan, and Oxaliplatin
  Other Names: Low doses of Gemcitabine; Low dose Fluorouracil [5FU]; Leucovorin; Low dose Irinotecan; Low dose Oxaliplatin)
Drug: G-FLIP-DM — G-FLIP-DM is low doses of Gemcitabine, Fluorouracil [5FU], Leucovorin, Irinotecan, Oxaliplatin, Docetaxel and Mitomycin C
  Other Names: Low dose Gemcitabine; Low dose Fluorouracil or 5FU; Leucovorin; Low dose Irinotecan; Low dose Oxaliplatin; Low dose Docetaxel; Low dose Mitomycin C
Dietary Supplement: Vitamin C — High dose of Vitamin C, used in combination with G-FLIP and then G-FLIP-DM
  Other Names: Ascorbic Acid
  Arms: G-FLIP+VitaminC, then G-FLIP-DM+VitaminC

SUMMARY:
Pancreatic cancer, especially at advanced metastatic stage, is a devastating disease. It is the fourth leading cause of cancer death. Its prognosis is grim - 5-year survival rate being 6%. The current therapies for advanced metastatic pancreatic cancer are very toxic and with limited efficacy. A safer and more effective therapy for this devastating disease is greatly needed.

G-FLIP regimen is a combination of low doses (doses lower than those approved by the FDA and used in the clinic) of several anti-cancer drugs, Gemcitabine, Fluorouracil, Leucovorin, Irinotecan and Oxaliplatin. The efficacy of G-FLIP against cancers (especially pancreatic cancer) is based on laboratory and clinical results, which indicates the synergistic efficacy of these anti-cancer drugs against cancer cells and overcoming tumor drug resistance that cancer cells frequently develop. Also, because of their low doses, this regimen is less toxic than when these drugs are used alone.

Meanwhile, intravenous infusion of high doses (doses significantly higher than the daily nutritional requirements) of Vitamin C (ascorbic acid) has been observed to have anti-cancer activities. This is especially true when Vitamin C is used in combination with other anti-cancer drugs.

DETAILED DESCRIPTION:
STUDY OBJECTIVE

The objective of this study is to evaluate the safety, tolerability and efficacy of G-FLIP (Low Doses of Gemcitabine, Fluorouracil [5FU], Leucovorin, Irinotecan, and Oxaliplatin), when used in combination with ascorbic acid (Vitamin C), as first-line therapy in patients with advanced pancreatic cancer. The objective of this study is also to evaluate the safety, tolerability and efficacy of G-FLIP-DM (G-FLIP + Low Doses of Docetaxel and Mitomycin C), when used in combination with ascorbic acid, in patients with advanced pancreatic cancer who develop Disease Progression (DP) with G-FLIP treatment. The primary endpoint is 12-month survival rate. The secondary endpoints include Overall Survival (OS), Quality of Life (QOL), Response Rate (RR), Progression-Free-Survival (PFS), and safety.

STUDY DRUGS

Study drugs include G-FLIP, G-FLIP-DM, and Vitamin C (Ascorbic Acid)

STUDY DESIGN

Sample Size:

There will be 34 "evaluable" study subjects in this study.

Treatments:

G-FLIP: All study subjects are treated with G-FLIP. Each treatment cycle of G-FLIP is 2 weeks, with G-FLIP given on Days 1 and 2 of each cycle. If study subjects exhibit Disease Progression (DP), treatment with G-FLIP will stop, and they will be treated with G-FLIP-DM.

G-FLIP-DM: Study subjects who exhibit DP with G-FLIP treatment will be treated with G-FLIP-DM. Each G-FLIP-DM treatment cycle is 2 weeks, with G-FLIP-DM given on Days 1 and 2 of each cycle.

Ascorbic Acid: Ascorbic acid will be administered twice weekly throughout the study, given on any 2 separate days of the week. Ascorbic acid will be administered throughout the study including during the follow-up period, even if treatment with G-FLIP or G-FLIP-DM has been terminated due to DP. Additionally, in 50% of the study subjects (i.e., 15 evaluable study subjects), treatment with ascorbic acid will begin on the same week when G-FLIP begins. In the other 50% of the study subjects (i.e., the other 15 evaluable study subjects), treatment with ascorbic acid will be delayed by 2 cycles. Results from these 2 groups of study subjects would allow comparison of potential acute safety of ascorbic acid, when used in combination with G-FLIP.

Open-Label: This is an open-label study, where investigators and study subjects are not blinded to the treatment.

Randomization: The assignment of study subjects will be randomized, as long as they meet eligibility criteria of the study.

DOSE DELAY AND DOSE MODIFICATION

In the event of adverse drug reactions, dose delay and dose modification will be dependent on the type of toxicities. The detailed dose modification scheme for G-FLIP, G-FLIP-DM and Ascorbic Acid are outlined in the protocol.

CONCOMITANT MEDICATIONS AND PROPHYLACTIC TREATMENT

Other than G-FLIP, G-FLIP-DM and ascorbic acid, patients cannot receive any other standard or investigational treatment for their cancer, or any study drugs for any non-cancer indications, while on this study. All concomitant medications (including names, dosage and schedule) must be recorded.

Prophylactic treatment for drug-related symptoms can be given according to Package Inserts of the study drugs and clinical practice. Supportive treatment may include anti-emetic, anti-diarrhea, anti-pyretic, anti-allergic, anti-hypertensive, analgesics, antibiotics, allopurinol, and others such as blood products and bone marrow growth factors. Patients may use erythropoietin for anemia. The investigator may utilize erythropoietic factors, or blood or platelet transfusions at their discretion.

DURATION OF TREATMENT AND FOLLOW-UP

At least six months of treatment is recommended for study subjects who have a response from G-FLIP or G-FLIP-DM, unless or until:

* Patients exhibit disease progression in the opinion of the principal investigator
* Unacceptable toxicity from the treatment
* Patient withdrawal of consent (Note: The investigator should make every effort to contact the subject to perform a final evaluation and to determine the reason(s) for withdrawal from the study.)
* Investigator's discretion to withdraw patients from the study because continued participation in the study is not in the patient's best interest.
* Underlying illness: a condition, injury, or disease unrelated to the intended disease which the study is investigating, that renders continuing treatment unsafe or regular follow-up impossible
* General or specific changes in the patient's condition that renders the patient ineligible for further investigational treatment
* Non-compliance with investigational treatment, protocol-required evaluations or follow-up visits

After treatment, study subjects should be followed so that information on survival and post study treatment are available for at least 1 year after the study subjects participate in the trial.

EFFICACY ASSESSMENTS

The efficacy of the study drugs will be assessed according to the following parameters:

Response Criteria of Complete Response (CR), Partial Response (PR), Stable Disease (SD), and Progressive Disease (Disease Progression or DP) will be derived from CT or MRI according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) (Eisenhauer et al. 2009).

Response Rate (RR) is the number of study subjects, expressed as a percentage of the total number of study subjects participated in the trial, who exhibit PR or CR that has been confirmed from 2 consecutive scans (CT or MRI).

Progression-Free-Survival (PFS) is the length of time when SD (or better) of a study subject is first documented until the time when DP, or death from any cause, occurs.

Overall Survival (OS) is the time from which the study subjects are first treated with G-FLIP to the time when death from any cause occurs. OS, which is the time from which the study subjects are first diagnosed with advanced pancreatic cancer to the time when death from any cause occurs, will also be recorded.

12-Month Survival Rate is the number of study subjects, expressed as a percentage of the total number of study subjects in the trial, who survive for 12 months starting from the time when the study subjects are accrued to the trial. The 12-Month Survival Rate for study subjects who survive for 12 months starting from the time when the study subjects are first diagnosed with advanced pancreatic cancer will also be recorded.

Safety Assessments

The efficacy of the study drugs will be assessed from the first dose to 1 month after last dose of the study drugs. The assessments will be based on the following parameters, performed at baselines and at various times during the study:

* physical exams
* evaluation of symptoms
* vital signs
* ECOG performance status and survival
* clinical pathology (clinical chemistry, renal function [assessed utilizing the Cockcroft-Gault formula], hematology, and coagulation)
* urinalysis
* QOL, assessed as described by Aaronson NK, et al. 1993.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically and cytologically confirmed metastatic (Stage IV), locally advanced unresectable (stage III), or locally recurrent pancreatic adenocarcinoma, with or without prior chemotherapy for their cancer.
* Eastern Cooperative Oncology Group (ECOG) performance status being 0-2.
* Expected survival >3 months.
* Patients 18 years of age and older of both genders.
* Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must use accepted contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive or double barrier device) during the study, and must have a negative serum or urine pregnancy test within 2 weeks prior to treatment initiation.
* Fertile men must practice effective contraceptive methods during the study, unless documentation of infertility exists.
* At least 2 weeks must have elapsed from any prior surgery or hormonal therapy.
* Laboratory values ≤2 weeks must be:

  * Adequate hematologic
  * Adequate hepatic function
  * Adequate renal function
* No evidence of active infection and no serious infections within the past month.
* Mentally competent, able to understand and willing to sign the informed consent form.

Exclusion Criteria:

* Patients under the age of 18.
* Locally advanced resectable disease from pancreatic cancer
* Previous radiotherapy for cerebral metastases, central nervous system (CNS) or epidural tumor.
* Patients receiving any other standard or investigational treatment for their cancer, or any other investigational agent for any non-cancer indication within the past 4 weeks.
* Patients with any active uncontrolled bleeding, or a bleeding diathesis.
* Pregnant women, or women of child-bearing potential not using reliable means of contraception.
* Lactating females.
* Fertile men unwilling to practice contraceptive methods during the study period.
* Life expectancy less than 3 months.
* Any condition or abnormality which may, in the opinion of the investigator, compromise the safety of patients.
* Unwilling or unable to follow protocol requirements.
* Active heart disease including but not limited to symptomatic congestive heart failure, symptomatic coronary artery disease, symptomatic angina pectoris, symptomatic myocardial infarction, or symptomatic congestive heart failure.
* Patients with a history of myocardial infarction that is < 3 months prior to registration.
* Patients with any amount of clinically significant pericardial effusion.
* Evidence of active serious infection.
* Patients with known HIV infection.
* Requirement for immediate palliative treatment of any kind including surgery and radiation.
* Patients that have received a chemotherapy regimen requiring stem cell support in the previous 6 months.
* Any condition or abnormality which may, in the opinion of the investigator, compromise the safety of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-08-13; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Azriel Hirschfeld, MD, Principal Investigator — Bruckner Oncology
Locations (1):
- Bruckner Oncology, The Bronx, New York, United States

REFERENCES:
- [Background] Bruckner H, Hirschfeld A, Buddaraju S, Stega J, Jahan M, Schwartz ME. Multidisciplinary effect of adding docetaxel and mitomycin-C to low-dose multidrug therapy for cholangiocarcinoma. J Clin Oncol 29: 2011 (suppl; abstr e14546)
- [Background] Bruckner HW, Myo M, Zaw K, Filipova O, Heidarian S, Rafiq N, Julliard K. Multi-drug chemotherapy for pancreatic cancer. Journal of Clinical Oncology 2005, 23 (16S. June 1 Supplement):4267 (abstract).
- [Background] Bruckner H, Simon K, Hrehorovich V. Low-dose sequential multi-drug regimens for advanced pancreatic cancer. Journal of Clinical Oncology, 2008, 26 (15S, May 20 Supplement) 15568 (Abstract)
- [Background] Monti DA, Mitchell E, Bazzan AJ, Littman S, Zabrecky G, Yeo CJ, Pillai MV, Newberg AB, Deshmukh S, Levine M. Phase I evaluation of intravenous ascorbic acid in combination with gemcitabine and erlotinib in patients with metastatic pancreatic cancer. PLoS One. 2012;7(1):e29794. doi: 10.1371/journal.pone.0029794. Epub 2012 Jan 17. PMID 22272248
- [Background] Goel A, Grossbard ML, Malamud S, Homel P, Dietrich M, Rodriguez T, Mirzoyev T, Kozuch P. Pooled efficacy analysis from a phase I-II study of biweekly irinotecan in combination with gemcitabine, 5-fluorouracil, leucovorin and cisplatin in patients with metastatic pancreatic cancer. Anticancer Drugs. 2007 Mar;18(3):263-71. doi: 10.1097/CAD.0b013e3280121334. PMID 17264757

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled: 13-August-2014;
  Last subject enrolled: 12-June-2017;
  Last investigational treatment: 21-June-2017.
Pre-assignment Details: Once consented, subjects were randomly assigned to one of the two arms, and then screened for eligibility.
Groups:
- G-FLIP + VitaminC, Then G-FLIP-DM + Vitamin C: G-FLIP in combination with Vitamin C were given. When Disease Progression occurred, G-FLIP-DM + Vitamin C were given.
  G-FLIP: G-FLIP is a combination of Low Doses of Gemcitabine, Fluorouracil [5FU], Leucovorin, Irinotecan, and Oxaliplatin
  G-FLIP-DM: G-FLIP-DM is low doses of Gemcitabine, Fluorouracil [5FU], Leucovorin, Irinotecan, Oxaliplatin, Docetaxel and Mitomycin C
  Vitamin C: High dose of Vitamin C, used in combination with G-FLIP and then G-FLIP-DM
- G-FLIP for 2 Weeks, Then G-FLIP + Vitamin C, Then G-FLIP-DM + Vitamin C: G-FLIP alone without Vitamin C for 2 weeks, then G-FLIP + Vitamin C. In the event of Disease Progression, G-GLIP-DM + Vitamin C were given.
  G-FLIP: G-FLIP is a combination of Low Doses of Gemcitabine, Fluorouracil [5FU], Leucovorin, Irinotecan, and Oxaliplatin
  G-FLIP-DM: G-FLIP-DM is low doses of Gemcitabine, Fluorouracil [5FU], Leucovorin, Irinotecan, Oxaliplatin, Docetaxel and Mitomycin C
Period: Overall Study
Arm/Group | G-FLIP + VitaminC, Then G-FLIP-DM + Vitamin C | G-FLIP for 2 Weeks, Then G-FLIP + Vitamin C, Then G-FLIP-DM + Vitamin C
Started (Disease Progrression) | 14 (Treatment was continued until study subjects exhibited Disease Progression with G-FLIP + Vitamin C, and until DP again with G-FLIP-DM + Vitamin C.) | 18 (Treatment was continued until study subjects exhibited Disease Progression with G-FLIP + Vitamin C, and until DP again with G-FLIP-DM + Vitamin C.)
Completed (Disease Progression) | 12 (Treatment was continued until study subjects exhibited Disease Progression with G-FLIP + Vitamin C, and until DP again with G-FLIP-DM + Vitamin C.) | 18 (Treatment was continued until study subjects exhibited Disease Progression with G-FLIP + Vitamin C, and until DP again with G-FLIP-DM + Vitamin C.)
Not Completed | 2 | 0
Not completed — Subjects was enrolled but did not start treatment because subjects have poor physical condition. | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- G-FLIP Alone for 4 Weeks, Then G-FLIP+VitaminC. When DP Occurred, Then G-FLIP-DM+VitaminC: G-FLIP in combination with Vitamin C. When Disease Progression occurred, then G-FLIP-DM + Vitamin C
  G-FLIP: G-FLIP is a combination of Low Doses of Gemcitabine, Fluorouracil [5FU], Leucovorin, Irinotecan, and Oxaliplatin
  G-FLIP-DM: G-FLIP-DM is low doses of Gemcitabine, Fluorouracil [5FU], Leucovorin, Irinotecan, Oxaliplatin, Docetaxel and Mitomycin C
  Vitamin C: High dose of Vitamin C, used in combination with G-FLIP and then G-FLIP-DM
- G-FLIP+VitaminC. When DP Occurred, Then G-FLIP-DM+Vitamin C.: G-FLIP alone for 2 weeks, then G-FLIP + Vitamin C. When Disease Progression occurred, then G-FLIP-DM + Vitamin C.
  G-FLIP: G-FLIP is a combination of Low Doses of Gemcitabine, Fluorouracil [5FU], Leucovorin, Irinotecan, and Oxaliplatin
  G-FLIP-DM: G-FLIP-DM is low doses of Gemcitabine, Fluorouracil [5FU], Leucovorin, Irinotecan, Oxaliplatin, Docetaxel and Mitomycin C
- Total: Total of all reporting groups
Arm/Group | G-FLIP Alone for 4 Weeks, Then G-FLIP+VitaminC. When DP Occurred, Then G-FLIP-DM+VitaminC | G-FLIP+VitaminC. When DP Occurred, Then G-FLIP-DM+Vitamin C. | Total
Number analyzed (Participants) | 14 | 18 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 12 | 17
  >=65 years | 9 | 6 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 10 | 12 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 18 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 14 | 17 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 18 | 32
Stage of Disease [Number; unit: participants] — Subjects must have Stage III or IV pancreatic cancer
  participants
    Stage III | 1 | 0 | 1
    Stage IV | 13 | 18 | 31

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Mean months subjects survived.
Time Frame: Survival was monitored from the first day of treatment until the date of death or last followed up.
Measure: Median (95% Confidence Interval); unit: Median months subjects survived
Arm/Group | G-FLIP Alone for 4 Weeks, Then G-FLIP+VitaminC. When DP Occurred, Then G-FLIP-DM+VitaminC | G-FLIP+VitaminC. When DP Occurred, Then G-FLIP-DM+Vitamin C.
Number analyzed (Participants) | 14 | 18
Median months subjects survived | 9.5 [2.5 to 19.3] | 10.1 [6.0 to 14.1]

2. Secondary Outcome: Objective Response
Description: Objective Response as a means of efficacy assessment was evaluated in terms of response rate. The response rate assessments included Complete Responses (CR), Partial Responses (PR), Overall Response Rate (ORR), Stable Disease (SD), and Disease Control Rate (DCR). The response rate was according to Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI. CR was disappearance of all target lesions. PR was >=30% decrease in the sum of the longest diameter of target lesions. ORR was CR + PR. SD was a condition that was not PR or Progressive Disease (PD). Finally, DCR was ORR + SD.
Time Frame: Performed before the start of treatment, at the beginning of each 2-week treatment cycle, at follow-up visit two weeks after completion of treatment, and for up to 3 years after the start of treatment.
Measure: Number; unit: Percentage
Arm/Group | G-FLIP Alone for 4 Weeks, Then G-FLIP+VitaminC. When DP Occurred, Then G-FLIP-DM+VitaminC | G-FLIP+VitaminC. When DP Occurred, Then G-FLIP-DM+Vitamin C.
Number analyzed (Participants) | 14 | 18
Percentage
  CR | 0.0 | 5.6
  PR | 14.3 | 33.3
  ORR | 14.3 | 38.9
  SD | 57.1 | 22.2
  DCR | 71.4 | 61.1

3. Other Pre Specified Outcome: Quality of Life Questionnaire
Description: Responses to Quality of Life questionnaire over a year since the start of treatment.
Time Frame: Performed before the start of treatment, at the beginning of each 2-week treatment cycle, and at follow-up visit two weeks after completion of treatment.
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Adverse Events
Description: The incidence of adverse events, as measured by blood tests, signs/symptoms, etc.
Time Frame: as for outcome 3
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Performed 1-2 weeks before the start of treatment, at the beginning of each 2-week treatment cycle, at follow-up visit two weeks after completion of treatment, and for up to 3 years.
Description: According to clinicaltrials.gov.
Arm/Group | G-FLIP Alone for 4 Weeks, Then G-FLIP+VitaminC. When DP Occurred, Then G-FLIP-DM+VitaminC | G-FLIP+VitaminC. When DP Occurred, Then G-FLIP-DM+Vitamin C.
All-Cause Mortality (participants affected / at risk) | 14/14 | 18/18
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/18
Other Adverse Events (participants affected / at risk) | 9/14 | 13/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | G-FLIP Alone for 4 Weeks, Then G-FLIP+VitaminC. When DP Occurred, Then G-FLIP-DM+VitaminC (N=14) | G-FLIP+VitaminC. When DP Occurred, Then G-FLIP-DM+Vitamin C. (N=18)
Anemia (Blood and lymphatic system disorders) | 1 | 2
Depression (Nervous system disorders) | 2 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 1
Fatigue (General disorders) | 2 | 2
Pain (General disorders) | 2 | 1
Insomnia (General disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 3 | 4
Anxiety (General disorders) | 2 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Anorexia (Blood and lymphatic system disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2015-01-06): https://cdn.clinicaltrials.gov/large-docs/50/NCT01905150/Prot_000.pdf
  • Statistical Analysis Plan (2015-01-06): https://cdn.clinicaltrials.gov/large-docs/50/NCT01905150/SAP_001.pdf